CLINICAL TRIAL: NCT04025554
Title: Anakinra for the Treatment of Chronically Inflamed White Matter Lesions in Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190124; 19-N-0124
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2023-10-25

CONDITIONS: Multiple Sclerosis
Keywords: Chronic Active Lesions; Ultra-high-field (7T) MRI; Interleukin-1 (IL-1); White Matter; Paramagnetic Rim
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1/Active treatment (Experimental): Patients with MS will be assigned to the same intervention
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — 100 mg daily weeks 1-4, 200 mg daily weeks 5-8, 300 mg daily weeks 9-12.

SUMMARY:
Background:

Multiple sclerosis (MS) is a disease of the central nervous system (CNS). People who have MS may have lesions that form on parts of the CNS, such as the brain. Some of these lesions may be inflamed for a long time. This causes MS to progress. There is no treatment for these lesions. Researchers believe that a drug that decreases inflammation can help.

Objective:

To see if a drug called anakinra can help clear inflammation in MS brain lesions.

Eligibility:

People 18 and older with MS and at least one white matter lesion.

Design:

Participants will be screened with one or more Neuroimmunology Clinic protocols.

Participants will have a medical history and physical exam. They will have blood and urine tests. They will have a lumbar puncture. For this, a needle is inserted between the bones in the back, and cerebrospinal fluid is removed. They will also have an MRI of the brain. The MRI scanner is a cylinder surrounded by a strong magnetic field. Participants will lie on a table that slides in and out of the scanner.

Participants will repeat the above procedures throughout the study.

Participants will get their first dose of anakinra at the clinic. They will administer the rest of the doses themselves, by injection under the skin.

Participants will track their daily dosage electronically or in a written drug diary.

Participants will have 4 visits while taking the drug. At each visit, sharps boxes and empty vials will be collected.

Participants will have 2 follow-up visits after completing treatment.

The study will last 28 weeks.

DETAILED DESCRIPTION:
Objective:

The overall goal of this study is to determine the safety, tolerability, and radiological efficacy of up to 12 weeks of subcutaneous injection of anakinra in people with multiple sclerosis and evidence, by magnetic resonance imaging (MRI), of chronic active (also known as smoldering ) lesions in the white matter.

Study population:

5 people with progressive or stable MS, at least one paramagnetic rim lesion on 7-tesla MRI, and no new white matter lesion formation for at least 3 months or clinical relapse for at least 12 months, will complete the study.

Design:

In this open label, dose escalation study, participants will receive up to 12 weeks of

subcutaneous anakinra with initial dose of 100 mg daily up to a target dose of 300 mg daily. Study visits will occur every 4 weeks while on treatment, with 2 follow-up visits at 4 and 12 weeks after treatment discontinuation.

Outcome measures:

The primary outcome measure is disappearance of one or more paramagnetic rims from white matter lesions identified at baseline. Secondary outcomes include safety and tolerability, clinical and radiological outcomes. Exploratory serological and CSF measures will also be obtained to investigate mechanism of action of anakinra and for biomarker development.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18
* Ability to give informed consent
* If fertile, agreement to use an effective method of birth control during the study and for up to 3 months after the last dose of the study drug
* Agreement not to participate in any other interventional study while participating in this protocol
* Diagnosis of MS, either stable or clinically progressive
* Prior 7-tesla MRI scan, with high image quality in the judgment of the study neuroradiologist, demonstrating at least one white matter lesion with a paramagnetic rim (41)

EXCLUSION CRITERIA:

* Pregnancy or current breastfeeding
* Use of another investigational agent within 1 month of screening
* Active infection and or neutropenia (ANC < 1000 cells/microliter)
* History of lymphoma
* Known hypersensitivity to administration of anakinra
* Previous treatment with anakinra and/or TNF-receptor inhibitor
* History of asthma
* QuantiFERON-TB gold positive
* Prior treatment with anti-CD20 agent (ocrelizumab, rituximab)
* Prior treatment with anti-CD52 agent (alemtuzumab)
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial or interfere with participation for the full duration of the trial; or not in the best interest of the subject to participate, in the opinion of the treating investigator
* Renal dysfunction, as defined by Clinical Center guidelines for administration of gadolinium
* Liver dysfunction, as indicated by baseline aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 1.5 times the upper limit of normal
* Clinical relapse in the 12 months prior to dosing
* New lesion formation (by comparison of screening MRI to a previous MRI of sufficient quality) in the 3 months prior to dosing
* One or more gadolinium-enhancing lesions on the screening scan
* Change in disease-modifying therapy in the 6 months prior to dosing
* Medical contraindication for 7-tesla MRI (including, but not limited to, any non-organic implant or other device such as a cardiac pacemaker or infusion pump or other metallic implants, objects, or body piercings, that are not MRI-compatible or cannot be removed)
* Psychological contraindication for 7-tesla MRI (e.g., claustrophobia)
* Contraindication to gadolinium administration.
* Active neoplastic disease or any medical condition, other than MS, that requires concurrent immunosuppression or immunomodulation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-N-0124.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled beginning on October 25, 2019 with the last participant enrolled on April 27, 2023. Candidates for participation were either 1) self referred, 2) referred by the Clinical Center Recruitment Office and NIH Clinical Research Volunteer Program or 3) identified during participation in an ongoing Neuroimmunology Clinic protocol.
Groups:
- All Participants: Participants with Multiple Sclerosis with at least one paramagnetic rim lesion noted on 7 Tesla MRI
Period: Overall Study
Arm/Group | All Participants
Started | 8
Completed | 5
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: Eight participants were treated with Anakinra. Three participants developed adverse events while on study drug. The study drug was discontinued and the three participants were withdrawn from the trial. The baseline characteristics include all participants who started on the study drug.
Groups:
- All Participants: Participants with Multiple Sclerosis with at least one paramagnetic rim lesion on 7T MRI, treated with Anakinra
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Modulation of One or All Paramagnetic Rim Lesions
Description: Proportion of lesions in which the paramagnetic rim has been modulated at the end of the dosing period.
Time Frame: 24 weeks
Measure: Number; unit: proportion of rim lesions modulated
Units Other Than Participants: Paramagnetic Rim Lesions
Groups:
- Treatment Group: Participants with Multiple Sclerosis with at least one paramagnetic rim lesion noted on 7 Tesla MRI, administered Anakinra starting at dose 100 mg/d up to a target dose of 300 mg/d
Arm/Group | Treatment Group
Number analyzed (Participants) | 5
Number analyzed (Paramagnetic Rim Lesions) | 25
proportion of rim lesions modulated | .04

2. Secondary Outcome: Change in the 9-hole Peg Test (9HPT)
Description: The Nine-Hole Peg Test (9-HPT) is a standardized, quantitative assessment used to measure finger dexterity. The test is administered by asking the participant to take pegs from a container, one by one, and place them into holes on a board as quickly as possible. Participants must then remove the pegs from the holes, one by one, and replace them back into the container. The test is timed with a lower number suggesting faster finger dexterity and a higher number suggesting slower finger dexterity. The results represent the mean change from baseline to end of dosing.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Treatment Group
Number analyzed (Participants) | 5
seconds | -0.42 (1.51)

3. Secondary Outcome: Change in the Symbol Digit Modalities Test (SDMT)
Description: The Symbol Digit Modalities Test (SDMT) is a neuropsychological test that assesses cognitive status, including processing speed, visual scanning, tracking, and motor speed. Participants are given a set of nine symbol-digit pairs and a sequence of symbols. They then have 90 seconds to match as many symbols in the sequence to their corresponding numbers as possible. The score is the number of correct substitutions within the 90 second interval, with a maximum of 110. The results represent a change from baseline to the end of dosing.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Treatment Group
Number analyzed (Participants) | 5
number correct | -3.6 (4.3)

4. Secondary Outcome: Change in the Expanded Disability Status Scale (EDSS)
Description: The EDSS is a tool used to measure the severity of multiple sclerosis (MS). The EDSS is based on a combination of scores from eight functional systems (FS), i.e., Muscle weakness, Balance, Coordination and Tremor, Eye Movements, Speech/Swallowing, Unusual Sensations or Numbness, Bowel and Bladder, Eyesight, and Thinking and Memory, and the Disability Status Scale (DSS). The EDSS is a scale that ranges from 0 to 10, with higher scores indicating greater disability. Scores of 1.0 to 4.5 indicate a high degree of ambulatory ability, while scores of 5.0 to 9.5 indicate a loss of ambulatory ability. The results represent a change from baseline to the end of dosing.
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: change in score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 5
change in score on a scale | 0 [0 to 0]

5. Secondary Outcome: Change in Paramagnetic Rim Lesion at Any Time Point
Description: Participants underwent 7T MRI during the dosing period and the post-dosing period. The results presented describe the proportion of paramagnetic rim lesions in which the rim was diminished or disappeared during the dosing period (weeks 0-12), during the post-dosing period (weeks 12-24) and during the entire study (weeks 0-24).
Time Frame: Up to 24 weeks
Measure: Median (Full Range); unit: Proportion of PRL changes
Units Other Than Participants: Paramagnetic Rim Lesions
Groups:
- Weeks 0-12: Proportion of paramagnetic rim lesions diminished or disappeared during the 0-12 week time period
- Weeks 12-24: Proportion of paramagnetic rim lesions diminished or disappeared during the 12-24 week time period
- Weeks 0-24: Proportion of paramagnetic rim lesions diminished or disappeared at any time during the 0-24 week time period
Arm/Group | Weeks 0-12 | Weeks 12-24 | Weeks 0-24
Number analyzed (Participants) | 5 | 5 | 5
Number analyzed (Paramagnetic Rim Lesions) | 25 | 21 | 21
Proportion of PRL changes | 0 [0 to 0.14] | 0 [0 to 0] | 0 [0 to 0.14]

6. Secondary Outcome: Change in Size of Paramagnetic Rim Lesions at All Time Points, Relative to Non-rim Lesions
Description: Paramagnetic rim lesions are multiple sclerosis plaques showing signs of low-grade, ongoing inflammation on MRI. Participants underwent MRI every 4 weeks and we compared the change in size between the participant's paramagnetic rim lesions (PRL+) and non-paramagnetic rim lesions (PRL-). At each time point, the mean group volume of each PRL+ and PRL- was calculated. The results provided include the group means and confidence limits at each time point for PRL+ and PRL- lesion type.
Time Frame: Every 4 weeks for the duration of the study
Measure: Geometric Mean (95% Confidence Interval); unit: mm^3
Units Other Than Participants: Lesions
Groups:
- PRL+: Paramagnetic Rim Lesions on 7T MRI
- PRL-: Non-Paramagnetic Rim Lesions noted on 7 Tesla MRI
Arm/Group | PRL+ | PRL-
Number analyzed (Participants) | 5 | 5
Number analyzed (Lesions) | 25 | 200
mm^3
  Baseline | 168.9 [114.4 to 252.8] | 50.7 [44.8 to 57.7]
  Week 4 | 168.4 [113.6 to 253.0] | 50.3 [44.4 to 57.2]
  Week 8 | 167.2 [112.6 to 251.8] | 49.9 [44.1 to 56.7]
  Week 12 | 175.4 [117.9 to 264.5] | 50.7 [44.8 to 57.7]
  Week 16 | 171.3 [115.9 to 256.4] | 46.9 [41.6 to 53.2]
  Week 24 | 160.5 [108.9 to 239.9] | 47.8 [42.4 to 54.3]

7. Secondary Outcome: Changes in T1 Relaxation Time Within Paramagnetic Rim Lesions at All Time Points, Relative to Non-rim Lesions
Description: Paramagnetic rim lesions are multiple sclerosis plaques showing signs of low-grade, ongoing inflammation on MRI. T1 relaxation time is a measure of brain damage on MRI. Participants underwent MRI every 4 weeks and we compared the change in T1 relaxation time between the participant's paramagnetic rim lesions (PRL+) and non-paramagnetic rim lesions (PRL-) at each time point. The results provided include the group means and confidence limits at each time point for PRL+ and PRL- lesion type.
Time Frame: Every 4 weeks for the duration of the study
Measure: Geometric Mean (95% Confidence Interval); unit: ms
Units Other Than Participants: Lesions
Groups:
- PRL+: Paramagnetic Rim Lesions noted on 7T MRI
- PRL-: Non-Paramagnetic Rim Lesions noted on 7T MRI
Arm/Group | PRL+ | PRL-
Number analyzed (Participants) | 5 | 5
Number analyzed (Lesions) | 25 | 200
ms
  Baseline | 1723 [1612 to 1858] | 1534 [1416 to 1697]
  Week 4 | 1708 [1599 to 1841] | 1522 [1407 to 1680]
  Week 8 | 1713 [1603 to 1848] | 1525 [1409 to 1683]
  Week 12 | 1706 [1597 to 1838] | 1522 [1407 to 1679]
  Week 16 | 1709 [1600 to 1841] | 1527 [1410 to 1687]
  Week 24 | 1728 [1616 to 1865] | 1525 [1409 to 1685]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of study participation, i.e., 24 weeks +/- 7 days.
Groups:
- All Participants: Participants with Multiple Sclerosis with at least one paramagnetic rim lesion on 7T MRI, administered Anakinra starting at dose 100 mg/d.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=8)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Injection site reaction (mild burning) (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Injection site reaction (erythema) (General disorders) | 5 (5)
Fatigue (General disorders) | 1 (1)
Injection site reaction (stinging) (General disorders) | 1 (2)
Injection site reaction (pruritus) (General disorders) | 3 (3)
Injection site reaction (edema) (General disorders) | 1 (1)
Injection site reaction (increased bleeding) (General disorders) | 1 (1)
Injection site reaction (pain) (General disorders) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders other specified; increased appetite (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - other; left achilles degenerative tendinosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Paresthesia (worsening) (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Nervous system disorder - other; hypoesthesia (middle dorsal lateral part of the feet) (Nervous system disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT04025554/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT04025554/ICF_001.pdf